CLINICAL TRIAL: NCT04379544
Title: Prognostic Value of Point of Care Cardiac and Lung Ultrasound in COVID-19
Acronym: CLUSCO
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 843008
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Coronavirus; Respiratory Failure
Keywords: COVID-19; Ultrasound; Point-of-care; Lung Ultrasound; Focused Echocardiography; Emergency Department; ICU
MeSH Terms: conditions — Coronavirus Infections; Respiratory Insufficiency; COVID-19; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 Positive Patients Receiving CPUS: Adult patients (18 years) presenting to the ED or ICU with highly suspected diagnosis or confirmed diagnosis of COVID-19 in whom the clinician deems a CPUS (cardiopulmonary ultrasound) is indicated.
  Interventions: Other: Observation only

INTERVENTIONS:
Other: Observation only — There is no intervention. This study is purely observational. This study simply follows COVID-19 patients who get CPUS based on their clinician deeming it necessary.

SUMMARY:
This is a protocol-driven observational study of lung ultrasound and focused echocardiography images obtained in the Emergency Department (ED) and Intensive Care Unit (ICU) settings as a part of existing standard of care. The objectives of this study are as follows:

1. To characterize various clinical and cardiopulmonary ultrasound findings and describe their relationship with the clinical course of patients with COVID-19 in the ED and ICU.
2. To describe, develop, and validate a prediction tool that can accurately predict the need for invasive mechanical ventilation (IMV) and acute respiratory failure in COVID-19 patients using clinical, laboratory, and ultrasound data.

DETAILED DESCRIPTION:
Background and scientific rationale:

During the COVID-19 pandemic, health care systems around the world are overwhelmed.

Surge of patients requiring hospital admission have led to shortages of ICU beds and mechanical ventilators. As an emerging clinical entity, little is known about the precise pathophysiologic mechanisms of COVID-19. Recent observational data and clinical experience has suggested that there could be different phenotypes of patients with COVID-19 which could explain the wide range of clinical presentations, response to therapies and outcomes.

Point of care cardiac and lung ultrasound (CLUS) has been proposed as a tool with potential to assist diagnostic evaluation and management of COVID-19 patients in the emergency department (ED) and intensive care unit (ICU) settings. Point of care CLUS is routinely used as part of the clinical evaluation of patients with dyspnea, hypoxemia, chest pain and shock in the ED and ICU. Patients with COVID-19 commonly present to the ED with these symptoms and therefore CLUS is being commonly used in patients with suspected or confirmed diagnosis of COVID-19.

Small observational studies have described several lung ultrasound (LUS) findings in patients with COVID-19. These findings include; pleural irregularity ("thickening"), subpleural consolidations, air bronchogram, isolated B-lines, fused B-lines and pleural effusions. Other observational studies have described the presence of acute myocardial abnormalities in patients with COVID-19 seen in echocardiography, including left and right ventricular systolic dysfunction.

Multiple studies have described and validated the finding of B-lines in LUS as a non-invasive marker of extravascular lung water. B-lines in LUS correlate with pulmonary capillary wedge pressures, NT-proBNP and E/e' and has been validated as a reliable prognostic factor in patients with decompensated heart failure. B-lines are also found in other pulmonary processes including viral pneumonia, ARDS, pulmonary contusions and post radiation changes. Observational studies involving COVID-19 patients have shown the presence of isolated and fused or continuous B-lines in the pneumonia associated with this infection. We hypothesize that the presence of B-lines in LUS may be marker of severity, and that alone or in concert with other clinical or laboratory variables, could help predict the clinical course and prognosis of COVID-19 patients.

Knowledge gaps

1. Does point of care cardiopulmonary ultrasound findings alone, or combined with other clinical and/or laboratory variables, predict clinical outcomes of patients with COVID-19?
2. Can different lung ultrasound finding patterns correlate with clinical severity or outcomes?

Specific aims

1. To characterize various clinical and CLUS findings and describe their relationship with clinical course of patients with COVID-19 in ED and ICU.
2. Using clinical, laboratory and ultrasound data to describe, develop and validate a prediction tool that can accurately predict (1) need of invasive mechanical ventilation (IVM) and (2) acute respiratory failure

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 positive or suspected positive
* Received a cardiopulmonary ultrasound scan

Exclusion Criteria:

* Did not receive a scan
* Not COVID-19 positive

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (>18 years) patients presenting to the ED and ICU with suspected diagnosis or confirmed diagnosis of COVID-19 in whom the clinician deems a CLUS indicated.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Patient requires invasive mechanical ventilation and suffers from acute respiratory failure. | 1 Year
  Number of patients requiring invasive mechanical ventilation and suffers from acute respiratory failure.
Patient is discharged | 1 Year
  Number of patients that do not require hospitalization and is able to safely recover from COVID-19 at home.
Patient is hospitalized, but does not require mechanical ventilation through the duration of hospital stay. | 1 Year
  Number of patients that must be hospitalized to recover from COVID-19, but does not require invasive mechanical ventilation and may or may not suffer from some degree of acute respiratory failure.

SECONDARY OUTCOMES:
Lung ultrasound findings | 1 year
  Any lung ultrasound findings including, but not limited to b-lines, a-lines, consolidations, pleural effusions and regularities. All of these findings are consolidated to a single score which will be the measure of the severity of lung ultrasound findings.
Cardiac ultrasound findings | 1 year
  Any cardiac ultrasound findings including, but not limited to IVC status, pericardial effusions, LV EF (%), RV function. All of these findings are consolidated to a single score which will be the measure of the severity of cardiac ultrasound findings.

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Teran, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Health System, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Grasselli G, Pesenti A, Cecconi M. Critical Care Utilization for the COVID-19 Outbreak in Lombardy, Italy: Early Experience and Forecast During an Emergency Response. JAMA. 2020 Apr 28;323(16):1545-1546. doi: 10.1001/jama.2020.4031. No abstract available. PMID 32167538
- [Background] Remuzzi A, Remuzzi G. COVID-19 and Italy: what next? Lancet. 2020 Apr 11;395(10231):1225-1228. doi: 10.1016/S0140-6736(20)30627-9. Epub 2020 Mar 13. PMID 32178769
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Background] Arentz M, Yim E, Klaff L, Lokhandwala S, Riedo FX, Chong M, Lee M. Characteristics and Outcomes of 21 Critically Ill Patients With COVID-19 in Washington State. JAMA. 2020 Apr 28;323(16):1612-1614. doi: 10.1001/jama.2020.4326. PMID 32191259
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Spencer KT, Kimura BJ, Korcarz CE, Pellikka PA, Rahko PS, Siegel RJ. Focused cardiac ultrasound: recommendations from the American Society of Echocardiography. J Am Soc Echocardiogr. 2013 Jun;26(6):567-81. doi: 10.1016/j.echo.2013.04.001. No abstract available. PMID 23711341
- [Background] Long B, Brady WJ, Koyfman A, Gottlieb M. Cardiovascular complications in COVID-19. Am J Emerg Med. 2020 Jul;38(7):1504-1507. doi: 10.1016/j.ajem.2020.04.048. Epub 2020 Apr 18. PMID 32317203
- [Background] Xie Y, Wang X, Yang P, Zhang S. COVID-19 Complicated by Acute Pulmonary Embolism. Radiol Cardiothorac Imaging. 2020 Mar 16;2(2):e200067. doi: 10.1148/ryct.2020200067. eCollection 2020 Apr. No abstract available. PMID 33778561
- [Background] Danzi GB, Loffi M, Galeazzi G, Gherbesi E. Acute pulmonary embolism and COVID-19 pneumonia: a random association? Eur Heart J. 2020 May 14;41(19):1858. doi: 10.1093/eurheartj/ehaa254. No abstract available. PMID 32227120
- [Background] Mitchell C, Collins K, Hua L, McClanahan C, Shea E, Umland M, Wasserman M. Specific Considerations for Sonographers When Performing Echocardiography during the 2019 Novel Coronavirus Outbreak: Supplement to the American Society of Echocardiography Statement. J Am Soc Echocardiogr. 2020 Jun;33(6):654-657. doi: 10.1016/j.echo.2020.04.014. Epub 2020 Apr 11. PMID 32503701
- [Background] Hendren NS, Drazner MH, Bozkurt B, Cooper LT Jr. Description and Proposed Management of the Acute COVID-19 Cardiovascular Syndrome. Circulation. 2020 Jun 9;141(23):1903-1914. doi: 10.1161/CIRCULATIONAHA.120.047349. Epub 2020 Apr 16. PMID 32297796
- [Background] Vieillard-Baron A, Price LC, Matthay MA. Acute cor pulmonale in ARDS. Intensive Care Med. 2013 Oct;39(10):1836-8. doi: 10.1007/s00134-013-3045-2. Epub 2013 Aug 2. No abstract available. PMID 23907498
- See also: Study information site — https://pennultrasound.org/clusco